CLINICAL TRIAL: NCT02307175
Title: A Phase I Study of 99m Tc Pertechnetate Produced in High Energy Cyclotron (CYCLOTEC) in Patients With Thyroid Scan Indication
Brief Title: A Study of 99m Tc Pertechnetate Produced in High Energy Cyclotron in Patients With Thyroid Scan Indication
Status: Completed | Type: Observational
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Dr Éric E Turcotte, MD, MD, Nuclear medicine specialist, Head of Clinical Research at CIMS, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Other Study IDs: CIMS-2014-01
Record Dates: First submitted 2014-09-24; First posted 2014-12-04 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Autoimmune Thyroid Disease; Congenital Hypothyroidism
MeSH Terms: conditions — Congenital Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cyclotec: The first 10 consecutively enrolled patients will have thyroid and whole body scan with CycloTec
- generator produced Tc99m-pertechnetate: 20 subsequent case-matched controls will have thyroid and whole body scan with conventional Tc99m-pertechnetate

SUMMARY:
Prospective, open label single site study to demonstrate the safety and efficacy of Tc-99m pertechnetate produced by high energy cyclotron at CHUS.

DETAILED DESCRIPTION:
The proposed clinical trial will be a prospective, case-controlled Phase I, open label, single site study. The first 10 consecutively enrolled patients will receive CYCLOTEC standard procedure thyroid imagery and an additional whole-body scans, and 20 subsequent case-matched controls, will receive GPERT and will also have additionnal whole body scan.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed thyroid scan
* Provided written informed consent prior to participation
* Biochemical parameters within 5 times of the normal limits for age
* WBC count > 3.0/μL
* ANC count 1.5/μL
* Platelets > 75,000/μL
* Haemoglobin > 10 g/dL
* Karnofsky Performance Scale score > 50

Exclusion Criteria:

* Nursing or pregnant females
* Biochemical parameters as measured outside 5 times the normal limits for age within 14 days of the scan
* WBC < 3.0/μL
* ANC < 1.5/μL
* Platelets < 75,000/μL
* Haemoglobin < 10 g/dL
* Unable and unwilling to follow instructions and comply with the protocol
* Unable or unwilling to provide written informed consent prior to participation in the study
* Karnofsky Performance Scale score < 50

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 80 years of age with thyroid scan indication
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Biodistribution of Tc99m produced by high-energy cyclotron (CycloTec) | 6 months
  Equivalence of biodistribution of Tc99m produced by high-energy cyclotron (CycloTec) will be compared to the biodistribution of the conventional Tc99m pertechnetated (Case match: 1 CycloTec patient vs. 2 conventional Tc99m-pertechnetate patients)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Turcotte, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada